CLINICAL TRIAL: NCT03139929
Title: Measurement of Mean Systemic Filling Pressure & Stressed Volume With CardioQ+® Oesophageal Doppler Measurement
Brief Title: Measurement of MSFP and Stressed Volume With CardioQ+®
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D.P.Veelo, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL 55531.018.15
Record Dates: First submitted 2017-04-03; First posted 2017-05-04 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cardiac Surgery; CABG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MSFP — MSFPhold and MSFParm

SUMMARY:
To study the reliablity of MSFP and stressed volume to follow volume loading and to predict fload loading responsiveness in patients after elective coronary artery bypass grafting (CABG) surgery.

DETAILED DESCRIPTION:
In this study the oesophageal Doppler monitor (CardioQ+), arterial pulse wave analysis (via the CardioQ+ and Flotrac device) and central venous pressure (CVP) will be used to estimate mean systemic filling pressure (MSFP) with the inspiratory hold method. Furthermore the MSFParm will be determined using a rapid cuff inflator. From MSFP vascular compliance (Csys) and stressed volume (Vs) will be calculated.

The accuracy of Vs to follow a 500 increase in volume will be studied. The accuracy of MSFP and Vs to to predict fluid loading responsiveness will be assessed in 42 patients after elective coronary artery bypass grafting (CABG) surgery. The effect of a standardised fluid loading on parameters of intrinsic contractility and afterload will be determined. The effect of fluid loading on inertia, resistance and elastance will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older planned for CABG

Exclusion Criteria:

* Contraindication for fluid loading
* Pregnancy, morbid obesity
* Hemodynamic instability with a mean arterial pressure (MAP) < 55 mm Hg and/ or a cardiac index < 1.5 L•min-1
* Severe arrhythmias
* Intra-cardiac shunts
* Symptomatic peripheral vascular disease
* Symptomatic pulmonary disease
* Significant valvular regurgitation
* Poor pre-operative left or right ventricular function
* Core temperature < 36 °C
* Contra-indication to the rapid cuff inflator
* Contra-indication to oesophageal Doppler probe insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CABG
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
MSFPhold | Before and after fluid administration (2 minutes and 10 minutes)
  Mean systemic filling pressure
MSFParm | Before and after fluid administration (2 minutes and 10 minutes)
  Mean systemic filling pressure

SECONDARY OUTCOMES:
Stressed volume | Before and after fluid administration (2 minutes and 10 minutes)
  Vs

OTHER OUTCOMES:
Vascular compliance (Csys) | Before and after fluid administration (2 minutes and 10 minutes)
  Vascular compliance
CVP | Before and after fluid administration (2 minutes and 10 minutes)
  central venous pressure
PPV | Before and after fluid administration (2 minutes and 10 minutes)
  pulse pressure variation
SVV | Before and after fluid administration (2 minutes and 10 minutes)
  stroke volume variation
Kinetic energy | Before and after fluid administration (2 minutes and 10 minutes)
  Kinetic energy

CONTACTS AND LOCATIONS:
Overall Officials: Bart Geerts, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijnberge M, Jansen JRC, Pinsky MR, Klanderman RB, Terwindt LE, Bosboom JJ, Lemmers N, Vlaar AP, Veelo DP, Geerts BF. Feasibility to estimate mean systemic filling pressure with inspiratory holds at the bedside. Front Physiol. 2022 Nov 29;13:1041730. doi: 10.3389/fphys.2022.1041730. eCollection 2022. PMID 36523553